CLINICAL TRIAL: NCT01702441
Title: Phase 1b/2a Open Label, Multiple-Ascending Dose Cohort Study to Assess the Safety, Tolerability, Pilot Efficacy, Pharmacokinetics and Pharmacodynamic Effects of 28 Day Repeat Subcutaneous Doses of AKB-9778 in Subjects With Diabetic Macular Edema
Brief Title: Safety and Pilot Efficacy of AKB-9778 in Subjects With Diabetic Macular Edema
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aerpio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKB-9778-CI-2002
Record Dates: First submitted 2012-09-24; First posted 2012-10-08 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Diabetic Macular Edema (DME)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AKB-9778 (Experimental): Up to 4 dose levels of subcutaneous AKB-9778 will be evaluated. Doses will be administered daily for 28 days.
  Interventions: Drug: Subcutaneous AKB-9778

INTERVENTIONS:
Drug: Subcutaneous AKB-9778

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, pharmacodynamics, and pilot efficacy of multiple ascending dose levels of AKB-9778 given as subcutaneous injections daily for 28 days in patients with diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

The following is an abbreviated list of inclusion criteria:

* Adults between 18 to 80 years of age, inclusive
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Decrease in vision determined to be primarily the result of DME in the study eye
* Definite Retinal thickening due to diffuse DME involving the center of the macula in the study eye
* Mean central subfield thickness of at least 325 µm by OCT in the study eye
* Early Treatment Diabetic Retinopathy Study (ETDRS) letter score BCVA ≤ 70 (20/40) in the study eye

Exclusion Criteria:

The following is an abbreviated list of exclusion criteria:

* Hemoglobin A1C (HbA1C) ≥ 11.5%
* History of any of the following in the study eye (however, the following are not exclusionary in the fellow eye):

  1. Panretinal scatter photocoagulation (PRP) or focal laser within 12 weeks prior to Screening
  2. Prior pars plana vitrectomy within 12 weeks prior to Screening
  3. Any ocular surgery within 12 weeks prior to Screening
  4. YAG capsulotomy within 7 days prior to Screening
  5. Prior intravitreal, subtenon, or periocular steroid therapy within 3 months prior to Screening or prior treatment with intravitreal anti-VEGF treatment within 1 month of Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs). | 28 days
Change from baseline in physical exams. | 28 days
Change from baseline in vital signs. | 28 days
Change from baseline in electrocardiograms (ECGs). | 28 days
Change from baseline in opthalmic exams. | 28 days
Change from baseline in clinical laboratory assay results. | 28 days
  Blood chemistry, hematology and urinalysis.

SECONDARY OUTCOMES:
Pharmacokinetics of AKB-9778 | Day 1 and Day 14
  Maximum plasma drug concentration (Cmax). Area under the plasma concentration-time curve (AUC).
Change from baseline in optical tomography (OCT)-measured retinal thickness. | 28 days
Change from baseline in best corrected visual acuity (BCVA). | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Peters, MD, Study Director — Aerpio Therapeutics
Locations (6):
- United States (6):
  - Beverly Hills, California
  - Winter Haven, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Charlotte, North Carolina
  - Cincinnati, Ohio